CLINICAL TRIAL: NCT01089556
Title: Use of Duloxetine or Pregabalin in Monotherapy Versus Combination Therapy of Both Drugs in Patients With Painful Diabetic Neuropathy "The COMBO - DN (COmbination vs Monotherapy of pregaBalin and dulOxetine in Diabetic Neuropathy) Study"
Brief Title: A Study in Painful Diabetic Neuropathy
Acronym: COMBO-DN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13084; F1J-EW-HMGQ (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-03-15; First posted 2010-03-18 (Estimated); Results first posted 2012-12-04 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Diabetic Neuropathy, Painful
MeSH Terms: conditions — Diabetic Neuropathies | interventions — Duloxetine Hydrochloride; Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Duloxetine (Experimental): Initial Treatment:
  Duloxetine 30 milligram (mg) daily for 1 week
  Duloxetine 60 mg daily for 7 weeks
  Intensive Treatment:
  Duloxetine 90 mg (60 mg in the morning, 30 mg in the evening) daily for 1 week
  Duloxetine 120 mg (60 mg twice daily) daily for 7 weeks
  Interventions: Drug: Duloxetine; Drug: Placebo
- Pregabalin+Duloxetine (Experimental): Initial Treatment:
  Pregabalin 150 mg daily for 1 week
  Pregabalin 300 mg (150 mg twice daily) daily for 7 weeks
  Intensive Treatment:
  Pregabalin 300 mg (150 mg twice daily) daily for 8 weeks
  Duloxetine 30 mg daily for 1 week
  Duloxetine 60 mg daily for 7 weeks
  Interventions: Drug: Duloxetine; Drug: Pregabalin; Drug: Placebo
- Pregabalin (Experimental): Initial Treatment:
  Pregabalin 150 mg daily for 1 week
  Pregabalin 300 mg (150 mg twice daily) daily for 7 weeks
  Intensive Treatment:
  Pregabalin 450 mg (300 mg in the morning, 150 mg in the evening) daily for 1 week
  Pregabalin 600 mg (300 mg twice daily) daily for 7 weeks
  Interventions: Drug: Pregabalin; Drug: Placebo
- Duloxetine + Pregabalin (Experimental): Initial Treatment:
  Duloxetine 30 mg daily for 1 week
  Duloxetine 60 mg daily for 7 weeks
  Intensive Treatment:
  Duloxetine 60 mg daily for 8 weeks
  Pregabalin 150 mg daily for 1 week
  Pregabalin 300 mg (150 mg twice daily) daily for 7 weeks
  Interventions: Drug: Duloxetine; Drug: Pregabalin; Drug: Placebo

INTERVENTIONS:
Drug: Duloxetine — Administered orally
  Other Names: Cymbalta; LY248686
  Arms: Duloxetine; Duloxetine + Pregabalin; Pregabalin+Duloxetine
Drug: Pregabalin — Administered orally
  Arms: Duloxetine + Pregabalin; Pregabalin; Pregabalin+Duloxetine
Drug: Placebo — Administered orally, daily as a blind for duloxetine and/or pregabalin for 8 or 16 weeks

SUMMARY:
This study will investigate the efficacy of a combination treatment of duloxetine + pregabalin compared with the maximal dose of each drug in monotherapy, in patients with diabetic peripheral neuropathic pain (DPNP) who have not responded to the standard recommended dose of either drug. It will provide an answer to a common clinical question, namely, is it better to increase the dose of the current monotherapy or to combine both treatments early on, in patients who do not respond to standard doses of duloxetine or pregabalin.

ELIGIBILITY:
Inclusion Criteria:

* Pain due to bilateral peripheral neuropathy (caused by type 1 or type 2 diabetes mellitus. Pain must begin in the feet, with relatively symmetrical onset. Daily pain should be present for more than 3 months [assessed by questioning patient]).
* Score of at least 4 on the 24-hour average pain severity score on an 11-point Likert scale [on Brief Pain Inventory (BPI) Modified Short Form] at screening and at randomization.
* Patient is currently not receiving treatment for diabetic peripheral neuropathic pain (DPNP) or was receiving treatment for DPNP, with a drug other than pregabalin or duloxetine, and completed the required washout
* Patient has never received treatment with duloxetine or pregabalin. (However, a short course of less than 15 days of treatment, at any time previously, will be allowed.)
* Stable glycemic control, as assessed by a physician investigator, and hemoglobin A1c (HbA1c) less than or equal to 12% at screening.

Exclusion Criteria:

* Have a known hypersensitivity to duloxetine or pregabalin or any of the inactive ingredients or have any contraindication for the use of duloxetine or pregabalin.
* Have uncontrolled narrow-angle glaucoma.
* Have received treatment with a monoamine oxidase inhibitor (MAOI) within 14 days prior to randomization, or have a potential need to use a MAOI during the study or within 5 days after discontinuation of study drug.
* Have received fluoxetine within 30 days prior to randomization.
* Have acute liver injury (such as hepatitis) or severe cirrhosis (Child-Pugh Class C).
* Have a serum creatinine greater than or equal to 1.5 milligram per deciliter (mg/dL) or a creatinine clearance less than 60 milliliter per minute (mL/min), at screening.
* Are judged clinically by the investigator to be at suicidal risk or as defined by a score of 2 or greater on Question 9 of the Beck Depression Inventory-II (BDI-II), at screening or randomization
* Have a historical exposure to drugs known to cause neuropathy (for example, vincristine), or a history of a medical condition, including pernicious anemia and hypothyroidism, that could have been responsible for neuropathy.
* Have pain that cannot be clearly differentiated from or conditions that interfere with the assessment of the DPNP.
* Have serious or unstable cardiovascular, hepatic, renal, respiratory or hematological illness; symptomatic peripheral vascular disease; a history of seizure disorder; or other medical (including unstable hypertension and not clinically euthyroid) or psychological conditions that, in the opinion of the investigator, would compromise participation or be likely to require hospitalization during the course of the study.
* Have received non-pharmacological treatment for pain within 14 days prior to randomization, or do not agree to abstain from non-pharmacological treatment during the study.
* Have a history of frequent and/or severe allergic reactions with multiple medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 811 (Actual)
Dates: Start 2010-03; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5AM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (54):
- Australia (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Newcastle, New South Wales
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Warrawong, New South Wales
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Elizabeth Vale, South Australia
- Canada (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kelowna, British Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vancouver, British Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Winnipeg, Manitoba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Halifax, Nova Scotia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cambridge, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Laval, Quebec
- Croatia (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Osijek
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rijeka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Varaždin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zagreb
- France (9):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Angers
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bourges
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Juan-les-Pins
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nevers
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nîmes
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Paris
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Valenciennes
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vierzon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vieux-Condé
- Germany (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dresden
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Schkeuditz
- Greece (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ampelokipoi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Athens
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Melíssia
- Italy (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Catania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Milan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Napoli
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rome
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mexico City, Mexico
- Netherlands (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Eindhoven
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Maastricht
- Poland (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bialystok
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lublin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Szczecin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wroclaw
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seoul, South Korea
- Spain (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Girona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Valencia
- Sweden (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Falköping
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Huddinge
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lund
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Stockholm
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zurich, Switzerland
- Turkey (Türkiye) (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ankara
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Izmir
- United Kingdom (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ashton-under-Lyne, Ashton-Under-Lyne
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chorley, Chorley
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Manchester, Greater Manchester
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ayrshire, Scotland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nuneaton, Warwickshire
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Livingston, West Lothian

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study consisted of 4 study periods (SP): 2 weeks screening and washout (SP I), 8 weeks initial treatment (SP II), 8 weeks intensive treatment (SP III), 2 weeks tapering (SP IV). Participants who did not achieve good pain control during SP II (<30% improvement) were considered non-responders and continued in the study and entered SP III.
Groups:
- Duloxetine (SP II): Duloxetine 30 milligram (mg) daily for Week 1 and 60 mg daily for Weeks 2-8 in Study Period II (SP II).
- Pregabalin (SP II): Pregabalin 150 mg daily for Week 1 and 300 mg daily for Weeks 2-8 in Study Period II.
- Duloxetine (SP III): Duloxetine 90 mg daily for Week 9 and 120 mg daily for Weeks 10-16 in Study Period III (SP III).
- DLX + PGB (SP III): Duloxetine (DLX) 60 mg plus Pregabalin (PGB) 150 mg daily for Week 9 and Duloxetine 60 mg plus Pregabalin 300 mg daily for Weeks 10-16 in Study Period III.
- PGB + DLX (SP III): Pregabalin (PGB) 300 mg plus Duloxetine (DLX) 30 mg daily for Week 9 and Pregabalin 300 mg plus Duloxetine 60 mg daily for Weeks 10-16 in Study Period III.
- Pregabalin (SP III): Pregabalin 450 mg daily for Week 9 and Pregabalin 600 mg daily for Weeks 10-16 in Study Period III.
Period: Study Period II (Weeks 1-8)
Arm/Group | Duloxetine (SP II) | Pregabalin (SP II) | Duloxetine (SP III) | DLX + PGB (SP III) | PGB + DLX (SP III) | Pregabalin (SP III)
Started | 404 | 407 | 0 | 0 | 0 | 0
Safety Population | 401 (Received at least 1 dose of study drug.) | 403 (Received at least 1 dose of study drug.) | 0 | 0 | 0 | 0
Non-responders Who Completed SPII | 158 | 205 | 0 | 0 | 0 | 0
Completed | 333 | 333 | 0 | 0 | 0 | 0
Not Completed | 71 | 74 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 35 | 39 | 0 | 0 | 0 | 0
Not completed — Entry Criteria Not Met | 12 | 8 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 1 | 2 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 3 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 4 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 4 | 4 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 12 | 14 | 0 | 0 | 0 | 0
Not completed — Not received any study drug | 3 | 4 | 0 | 0 | 0 | 0
Period: Study Period III (Weeks 9-16)
Arm/Group | Duloxetine (SP II) | Pregabalin (SP II) | Duloxetine (SP III) | DLX + PGB (SP III) | PGB + DLX (SP III) | Pregabalin (SP III)
Started | 0 | 0 | 74 (Of those who completed SPII, 10 non-responders did not enter SPIII, while 4 responders entered SPIII) | 75 (Of those who completed SPII, 6 non-responders did not enter SPIII, while 3 responders entered SPIII) | 95 (Of those who completed SPII, 10 non-responders did not enter SPIII, while 4 responders entered SPIII) | 99 (Of those who completed SPII, 6 non-responders did not enter SPIII, while 1 responders entered SPIII)
Efficacy and Safety Population | 0 | 0 | 73 (Received ≥1 dose study drug, had Week 8 and at least 1 assessment during Weeks 9-16 (SPIII)) | 75 (Received ≥1 dose study drug, had Week 8 and at least 1 assessment during Weeks 9-16 (SPIII)) | 94 (Received ≥1 dose study drug, had Week 8 and at least 1 assessment during Weeks 9-16 (SPIII)) | 97 (Received ≥1 dose study drug, had Week 8 and at least 1 assessment during Weeks 9-16 (SPIII))
Completed | 0 | 0 | 60 | 66 | 83 | 92
Not Completed | 0 | 0 | 14 | 9 | 12 | 7
Not completed — Adverse Event | 0 | 0 | 4 | 2 | 4 | 3
Not completed — Entry Criteria Not Met | 0 | 0 | 1 | 1 | 1 | 1
Not completed — Lack of Efficacy | 0 | 0 | 0 | 2 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 1 | 1 | 0
Not completed — Satisfactory Response | 0 | 0 | 4 | 3 | 4 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 3 | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Duloxetine: Duloxetine 30 milligram (mg) daily for Week 1 and 60 mg daily for Weeks 2-8 in Study Period II.
- Pregabalin: Pregabalin 150 mg daily for Week 1 and 300 mg daily for Weeks 2-8 in Study Period II.
- Total: Total of all reporting groups
Arm/Group | Duloxetine | Pregabalin | Total
Number analyzed (Participants) | 401 | 403 | 804
Age Continuous [Mean (Standard Deviation); unit: years] | 61.5 (10.62) | 61.9 (10.95) | 61.7 (10.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 182 | 174 | 356
  Male | 219 | 229 | 448
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 37 | 36 | 73
  Asian | 34 | 34 | 68
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 2 | 2 | 4
  White | 324 | 328 | 652
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 3 | 6
Region of Enrollment [Number; unit: participants]
  Greece | 16 | 12 | 28
  Spain | 6 | 8 | 14
  Turkey | 5 | 7 | 12
  United Kingdom | 31 | 31 | 62
  Italy | 16 | 18 | 34
  France | 22 | 24 | 46
  Mexico | 75 | 71 | 146
  Canada | 19 | 19 | 38
  Poland | 56 | 57 | 113
  Croatia | 27 | 29 | 56
  Australia | 27 | 22 | 49
  Netherlands | 5 | 4 | 9
  Germany | 52 | 54 | 106
  Korea, Republic of | 31 | 32 | 63
  Sweden | 13 | 15 | 28
Clinical Global Impressions of Severity Scale (CGI-S) [Mean (Standard Deviation); unit: units on a scale] — The clinician recorded how ill the participant was at the time of assessment, in relation to the clinician's total experience with this participant population. Scores range from 1 (normal, not at all ill) to 7 (among the most extremely ill participants). One participant in Duloxetine group and 2 participants in Pregabalin group had missing data and were not included in the calculation of mean and standard deviation (SD).
  units on a scale | 4.0 (1.07) | 4.0 (1.09) | 4.0 (1.08)
Patient Global Impressions of Severity Scale (PGI-S) [Mean (Standard Deviation); unit: units on a scale] — Measures participant's perception of severity of illness at the time of assessment. Scores range from 1 (normal, not at all ill) to 7 (extremely ill).
  units on a scale | 3.4 (1.42) | 3.4 (1.41) | 3.4 (1.42)
Brief Pain Inventory (BPI) Severity: Average Pain Score [Mean (Standard Deviation); unit: units on a scale] — A self-reported scale that measures the severity of pain based on the average pain experienced over the past 24-hours. The severity scores range from 0 (no pain) to 10 (pain as severe as you can imagine). Two participants in Pregabalin group had missing data and were not included in the calculation of mean and SD.
  units on a scale | 6.0 (1.55) | 6.0 (1.57) | 6.0 (1.56)
Neuropathic Pain Symptom Inventory (NPSI) [Mean (Standard Deviation); unit: units on a scale] — The NPSI is a 12-item self-administered questionnaire to assess 5 different dimensions of neuropathic pain: superficial spontaneous burning pain, deep spontaneous pressing pain, paroxysmal pain, evoked pains, and paresthesias/dysesthesias. Questionnaire generates a score in each of the relevant dimensions and a total score of 0-100. Higher score indicates a greater intensity of pain. Two participants in Duloxetine group and 6 participants in Pregabalin group had missing data and were not included in the calculation of mean and SD.
  units on a scale | 47.3 (19.16) | 47.7 (20.46) | 47.5 (19.81)
Hospital Anxiety and Depression Scale (HADS) - Anxiety Subscale Score [Mean (Standard Deviation); unit: units on a scale] — A 14-item questionnaire with 2 subscales: anxiety and depression. Each item is rated on a 4-point scale (0-3), giving maximum scores of 21 for anxiety and for depression. Scores of 11 or more on either subscale are considered to be a significant case of psychological morbidity, while scores of 8-10 represent 'borderline' and 0-7, 'normal.' Three participants in both Duloxetine group and Pregabalin group had missing data and were not included in the calculation of mean and SD.
  units on a scale | 6.8 (4.31) | 6.6 (4.32) | 6.7 (4.31)
Hospital Anxiety and Depression Scale (HADS) - Depression Subscale Score [Mean (Standard Deviation); unit: units on a scale] — A 14-item questionnaire with 2 subscales: anxiety and depression. Each item is rated on a 4-point scale (0-3), giving maximum scores of 21 for anxiety and for depression. Scores of 11 or more on either subscale are considered to be a significant case of psychological morbidity, while scores of 8-10 represent 'borderline' and 0-7, 'normal.' Two participants in Duloxetine group and 1 participant in Pregabalin group had missing data and were not included in the calculation of mean and SD.
  units on a scale | 5.5 (4.19) | 5.5 (3.88) | 5.5 (4.04)
Sheehan Disability Scale (SDS) [Mean (Standard Deviation); unit: units on a scale] — The SDS is completed by the participants and is used to assess the effect of their symptoms on work (Item 1), social (Item 2) and family life (Item 3). Each item is measured on a 0 (not at all) to 10 (extremely) point scale with higher values indicating greater disruption. Total scores is the sum of the 3 items and range from 0-30 with higher values indicating greater disruption in the participant's work/social/family life. There were 118 participants in Duloxetine group and 128 participants in Pregabalin group who had missing data and were not included in the calculation of mean and SD.
  units on a scale | 13.3 (7.47) | 13.3 (7.59) | 13.3 (7.52)
Average number of hours worked for pay per week [Mean (Standard Deviation); unit: hours] — Data presented are average number of hours worked for pay per week during last 8 weeks prior to entering Study Period II. There were 275 participants in Duloxetine group and 281 participants in Pregabalin group who had missing data and were not included in the calculation of mean and SD.
  hours | 39.5 (20.33) | 41.4 (16.36) | 40.4 (18.47)
Number of days of work/school missed [Mean (Standard Deviation); unit: days] — Data presented are the number of days of work/school missed due to diabetic peripheral neuropathic pain (DPNP) during the last 8 weeks prior to entering Study Period II. There were 278 participants in Duloxetine group and 281 participants in Pregabalin group who had missing data and were not included in the calculation of mean and SD.
  days | 2.3 (7.98) | 1.3 (4.69) | 1.8 (6.56)
Number of days hospitalized [Mean (Standard Deviation); unit: days] — Data presented are the number of days hospitalized due to DPNP during the last 8 weeks prior to entering Study Period II. There were 21 participants in Duloxetine group and 23 participants in Pregabalin group who had missing data and were not included in the calculation of mean and SD.
  days | 0.0 (0.45) | 0.1 (0.67) | 0.1 (0.57)
Blood pressure (BP) [Mean (Standard Deviation); unit: millimeter of mercury (mm Hg)] — One participant in both Duloxetine group and Pregabalin group had missing data and were not included in the calculation of mean and SD.
  millimeter of mercury (mm Hg)
    Systolic BP | 135.0 (16.27) | 134.3 (15.62) | 134.7 (15.94)
    Diastolic BP | 77.6 (10.04) | 76.7 (9.43) | 77.1 (9.74)
Pulse rate [Mean (Standard Deviation); unit: beats per minute (bpm)] — Three participants in Duloxetine group and 1 participant in Pregabalin group had missing data and were not included in the calculation of mean and SD.
  beats per minute (bpm) | 76.0 (10.81) | 75.6 (11.05) | 75.8 (10.92)

OUTCOME MEASURES:

1. Primary Outcome: Change From Week 8 to Week 16 Endpoint in 24 Hour Average Pain Item Score on the Brief Pain Inventory (BPI) Modified Short Form
Description: BPI Modified Short Form 24-Hour average pain item score is a self-reported scale that measures the severity of pain based on the average pain experienced over the past 24 hours. The severity scores range from 0 (no pain) to 10 (pain as severe as you can imagine). Mixed-effects model repeated measures (MMRM) analysis was used to calculate Least Squares (LS) Mean and 95% Confidence Interval (CI). LS Mean values are controlled for treatment, site, baseline value, visit, treatment*visit, baseline*visit and treatment in Study Period II.
Time Frame: Week 8, Week 16
Population: All randomized participants who received at least one dose of study drug, and had Week 8 and at least one BPI measurements during Weeks 9-16 (Study Period III).
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Combination: All participants who received Duloxetine Combination therapy (Duloxetine 60 milligram [mg] plus Pregabalin 150 mg daily for Week 9 and Duloxetine 60 mg plus Pregabalin 300 mg daily for Weeks 10-16) or Pregabalin Combination therapy (Pregabalin 300 mg plus Duloxetine 30 mg daily for Week 9 and Pregabalin 300 mg plus Duloxetine 60 mg daily for Weeks 10-16) in Study Period III were pooled together.
- Monotherapy: All participants who received Duloxetine Monotherapy (Duloxetine 90 mg daily for Week 9 and 120 mg daily for Weeks 10-16) or Pregabalin Monotherapy (Pregabalin 450 mg daily for Week 9 and Pregabalin 600 mg daily for Weeks 10-16) in Study Period III were pooled together.
Arm/Group | Combination | Monotherapy
Number analyzed (Participants) | 169 | 170
units on a scale | -2.353 [-2.688 to -2.017] | -2.161 [-2.509 to -1.812]
Statistical Analysis 1: Comparison: Combination vs Monotherapy; Test type: Superiority or Other; p = 0.370, Mixed Models Analysis; LS Mean Differences (Final Values) = -0.192

2. Other Pre Specified Outcome: Mean Change From Baseline to Week 8 Endpoint in 24 Hour Average Pain Item Score on the Brief Pain Inventory (BPI) Modified Short Form
Description: BPI Modified Short Form 24-Hour average pain item score is a self-reported scale that measures the severity of pain based on the average pain experienced over the past 24 hours. The severity scores range from 0 (no pain) to 10 (pain as severe as you can imagine). Mixed-effects model repeated measures (MMRM) analysis was used to calculate Least Squares (LS) Mean and 95% Confidence Interval (CI). LS Mean values are controlled for treatment, site, baseline value, visit, treatment*visit and baseline*visit.
Time Frame: Baseline, Week 8
Population: All randomized participants who received at least one dose of study drug, and had baseline and at least one post-baseline BPI measurements during Weeks 1-8 (Study Period II).
Measure: Least Squares Mean (90% Confidence Interval); unit: units on a scale
Arm/Group | Duloxetine | Pregabalin
Number analyzed (Participants) | 401 | 401
units on a scale | -2.295 [-2.508 to -2.083] | -1.682 [-1.893 to -1.471]
Statistical Analysis 1: Comparison: Duloxetine vs Pregabalin; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; LS Mean Differences (Final Values) = -0.614

3. Secondary Outcome: Mean Change From Week 8 to Week 16 Endpoint in Items of the Brief Pain Inventory (BPI) Modified Short Form Worst Pain Score
Description: BPI Modified Short Form worst pain score is a self-reported scale that measures the severity of pain based on the worst pain experienced over the past 24 hours. The severity scores range from 0 (no pain) to 10 (pain as severe as you can imagine). Mixed-effects model repeated measures (MMRM) analysis was used to calculate Least Squares (LS) Mean and 95% Confidence Interval (CI). LS Mean values are controlled for treatment, site, baseline value, visit, treatment*visit, baseline*visit and treatment in Study Period II.
Time Frame: Week 8, Week 16
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Combination | Monotherapy
Number analyzed (Participants) | 169 | 170
units on a scale | -2.374 [-2.757 to -1.990] | -2.371 [-2.771 to -1.971]
Statistical Analysis 1: Comparison: Combination vs Monotherapy; Test type: Superiority or Other; p = 0.991, Mixed Models Analysis; LS Mean Differences (Final Values) = -0.003

4. Other Pre Specified Outcome: Percentage of Participants With a Reduction of Greater Than or Equal to 30% on Brief Pain Inventory (BPI) Modified Short Form 24-Hour Average Pain Item Score at Week 8 Endpoint
Description: BPI Modified Short Form 24-Hour average pain item score is a self-reported scale that measures the severity of pain based on the average pain experienced over the past 24 hours. The severity scores range from 0 (no pain) to 10 (pain as severe as you can imagine).
Time Frame: Baseline through Week 8
Population: All randomized participants who received at least one dose of study drug, and had baseline and at least one post-baseline BPI measurements during Weeks 1-8 (Study Period II). Last observation carried forward (LOCF) principle was used.
Measure: Number; unit: percentage of participants
Arm/Group | Duloxetine | Pregabalin
Number analyzed (Participants) | 375 | 374
percentage of participants | 52.0 | 36.9
Statistical Analysis 1: Comparison: Duloxetine vs Pregabalin; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 1.431, 95% CI 2-sided [1.233 to 1.662]

5. Secondary Outcome: Percentage of Participants With a Reduction of Greater Than or Equal to 30% on Brief Pain Inventory (BPI) Modified Short Form 24-Hour Average Pain Item Score at Week 16 Endpoint
Description: as for outcome 4
Time Frame: Week 8 through Week 16
Population: All randomized participants who received at least one dose of study drug, and had Week 8 and at least one BPI measurements during Weeks 9-16 (Study Period III). Last observation carried forward (LOCF) principle was used.
Measure: Number; unit: percentage of participants
Arm/Group | Combination | Monotherapy
Number analyzed (Participants) | 165 | 163
percentage of participants | 61.8 | 55.8
Statistical Analysis 1: Comparison: Combination vs Monotherapy; Test type: Superiority or Other; p = 0.565, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 1.052, 95% CI 2-sided [0.884 to 1.253]

6. Other Pre Specified Outcome: Percentage of Participants With a Reduction of Greater Than or Equal to 50% on Brief Pain Inventory (BPI) Modified Short Form 24-Hour Average Pain Item Score at Week 8 Endpoint
Description: as for outcome 4
Time Frame: Baseline through Week 8
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Duloxetine | Pregabalin
Number analyzed (Participants) | 375 | 374
percentage of participants | 40.3 | 27.8
Statistical Analysis 1: Comparison: Duloxetine vs Pregabalin; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 1.467, 95% CI 2-sided [1.214 to 1.771]

7. Secondary Outcome: Percentage of Participants With a Reduction of Greater Than or Equal to 50% on Brief Pain Inventory (BPI) Modified Short Form 24-Hour Average Pain Item Score at Week 16 Endpoint
Description: as for outcome 4
Time Frame: Week 8 through Week 16
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Combination | Monotherapy
Number analyzed (Participants) | 165 | 163
percentage of participants | 52.1 | 39.3
Statistical Analysis 1: Comparison: Combination vs Monotherapy; Test type: Superiority or Other; p = 0.068, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 1.233, 95% CI 2-sided [0.980 to 1.550]

8. Other Pre Specified Outcome: Percentage of Participants With a Decrease of Greater Than or Equal to 2 Points on Brief Pain Inventory (BPI) Modified Short Form 24-Hour Average Pain Item Score at Week 8 Endpoint
Description: as for outcome 4
Time Frame: Baseline through Week 8
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Duloxetine | Pregabalin
Number analyzed (Participants) | 375 | 374
percentage of participants | 57.1 | 45.7
Statistical Analysis 1: Comparison: Duloxetine vs Pregabalin; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 1.279, 95% CI 2-sided [1.125 to 1.456]

9. Secondary Outcome: Percentage of Participants With a Decrease of Greater Than or Equal to 2 Points on Brief Pain Inventory (BPI) Modified Short Form 24-Hour Average Pain Item Score at Week 16 Endpoint
Description: as for outcome 4
Time Frame: Week 8 through Week 16
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Combination | Monotherapy
Number analyzed (Participants) | 165 | 163
percentage of participants | 66.7 | 64.4
Statistical Analysis 1: Comparison: Combination vs Monotherapy; Test type: Superiority or Other; p = 0.843, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 0.985, 95% CI 2-sided [0.842 to 1.151]

10. Other Pre Specified Outcome: Clinical Global Impression of Improvement (CGI-I) at Week 8 Endpoint
Description: Measures clinician's perception of participant improvement at the time of assessment compared with the start of treatment. Scores range from 1 (very much better) to 7 (very much worse). Mixed-effects model repeated measures (MMRM) analysis was used to calculate Least Squares (LS) Mean and 95% Confidence Interval (CI). LS Mean values are controlled for treatment, site, visit, and treatment*visit.
Time Frame: Week 8
Population: All randomized participants who received at least one dose of study drug, and had at least one post-baseline CGI-I measurement during Weeks 1-8 (Study Period II).
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Duloxetine | Pregabalin
Number analyzed (Participants) | 400 | 401
units on a scale | 2.508 [2.396 to 2.619] | 2.848 [2.737 to 2.959]
Statistical Analysis 1: Comparison: Duloxetine vs Pregabalin; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; LS Mean Difference (Final Values) = -0.341

11. Secondary Outcome: Clinical Global Impression of Improvement (CGI-I) at Week 16 Endpoint
Description: Measures clinician's perception of participant improvement at the time of assessment compared with the start of treatment for Study Period III. Scores range from 1 (very much better) to 7 (very much worse). Mixed-effects model repeated measures (MMRM) analysis was used to calculate Least Squares (LS) Mean and 95% Confidence Interval (CI). LS Mean values are controlled for treatment, site, baseline value, visit, treatment*visit, baseline*visit and treatment in Study Period II.
Time Frame: Week 16
Population: All randomized participants who received at least one dose of study drug, and had at least one CGI-I measurement during Weeks 9-16 (Study Period III).
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Combination | Monotherapy
Number analyzed (Participants) | 169 | 170
units on a scale | 2.286 [2.127 to 2.444] | 2.359 [2.193 to 2.524]
Statistical Analysis 1: Comparison: Combination vs Monotherapy; Test type: Superiority or Other; p = 0.475, Mixed Models Analysis; LS Mean Difference (Final Values) = -0.073

12. Other Pre Specified Outcome: Mean Change From Baseline to Week 8 Endpoint on the Neuropathic Pain Symptom Inventory (NPSI) Questionnaire
Description: The NPSI is a 12-item self-administered questionnaire to assess 5 different dimensions of neuropathic pain: superficial spontaneous burning pain, deep spontaneous pressing pain, paroxysmal pain, evoked pains, and paresthesias/dysesthesias. A total score ranges from 0 to 100. Higher score indicates a greater intensity of pain. Mixed-effects model repeated measures (MMRM) analysis was used to calculate Least Squares (LS) Mean and 95% Confidence Interval (CI). LS Mean values are controlled for treatment, site, baseline value, visit, treatment*visit and baseline*visit.
Time Frame: Baseline, Week 8
Population: All randomized participants who received at least one dose of study drug, and had baseline and at least one post-baseline NPSI measurements during Weeks 1-8 (Study Period II).
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Duloxetine | Pregabalin
Number analyzed (Participants) | 399 | 397
units on a scale | -19.442 [-21.366 to -17.518] | -14.684 [-16.606 to -12.762]
Statistical Analysis 1: Comparison: Duloxetine vs Pregabalin; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; LS Mean Difference (Final Values) = -4.758

13. Secondary Outcome: Mean Change From Week 8 to Week 16 Endpoint on the Neuropathic Pain Symptom Inventory (NPSI) Questionnaire
Description: The NPSI is a 12-item self-administered questionnaire to assess 5 different dimensions of neuropathic pain: superficial spontaneous burning pain, deep spontaneous pressing pain, paroxysmal pain, evoked pains, and paresthesias/dysesthesias. A total score ranges from 0 to 100. Higher score indicates a greater intensity of pain. Mixed-effects model repeated measures (MMRM) analysis was used to calculate Least Squares (LS) Mean and 95% Confidence Interval (CI). LS Mean values are controlled for treatment, site, baseline value, visit, treatment*visit, baseline*visit and treatment in Study Period II.
Time Frame: Week 8, Week 16
Population: All randomized participants who received at least one dose of study drug, and had Week 8 and at least one NPSI measurements during Weeks 9-16 (Study Period III).
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Combination | Monotherapy
Number analyzed (Participants) | 169 | 170
units on a scale | -13.734 [-16.588 to -10.880] | -11.801 [-14.774 to -8.828]
Statistical Analysis 1: Comparison: Combination vs Monotherapy; Test type: Superiority or Other; p = 0.289, Mixed Models Analysis; LS Mean Difference (Final Values) = -1.933

14. Other Pre Specified Outcome: Mean Change From Baseline to Week 8 Endpoint in Sheehan Disability Scale (SDS)
Description: The SDS is completed by the participant and is used to assess the effect of the participant's symptoms on their work (Item 1), social (Item 2), and family life (Item 3). Each item is measured on a 0 (not at all) to 10 (extremely) point scale with higher values indicating greater disruption. Total scores is the sum of the 3 items and range from 0 to 30 with higher values indicating greater disruption in the participant's work/social/family life. Least Squares (LS) mean values are controlled for treatment, site, baseline value and treatment*site.
Time Frame: Baseline, Week 8
Population: All randomized participants who received at least one dose of study drug, and had baseline and at least one post-baseline SDS measurement during Weeks 1-8 (Study Period II). Last observation carried forward (LOCF) principle was used.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Duloxetine | Pregabalin
Number analyzed (Participants) | 235 | 234
units on a scale | -4.387 [-5.185 to -3.590] | -3.367 [-4.133 to -2.601]
Statistical Analysis 1: Comparison: Duloxetine vs Pregabalin; Test type: Superiority or Other; p = 0.071, ANCOVA; LS Mean Difference (Final Values) = -1.020

15. Secondary Outcome: Mean Change From Week 8 to Week 16 Endpoint in Sheehan Disability Scale (SDS)
Description: The SDS is completed by the participant and is used to assess the effect of the participant's symptoms on their work (Item 1), social (Item 2), and family life (Item 3). Each item is measured on a 0 (not at all) to 10 (extremely) point scale with higher values indicating greater disruption. Total scores is the sum of the 3 items and range from 0 to 30 with higher values indicating greater disruption in the participant's work/social/family life. Least Squares (LS) Mean values are controlled for treatment, site, baseline value, treatment*site and treatment in Study Period II.
Time Frame: Week 8, Week 16
Population: All randomized participants who received at least one dose of study drug, and had Week 8 and at least one SDS measurement during Weeks 9-16 (Study Period III). Last observation carried forward (LOCF) principle was used.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Combination | Monotherapy
Number analyzed (Participants) | 108 | 106
units on a scale | -2.625 [-3.589 to -1.661] | -2.431 [-3.410 to -1.453]
Statistical Analysis 1: Comparison: Combination vs Monotherapy; Test type: Superiority or Other; p = 0.780, ANCOVA; LS Mean Difference (Final Values) = -0.193

16. Other Pre Specified Outcome: Mean Change From Baseline to Week 8 Endpoint in Hospital Anxiety and Depression Scale (HADS)
Description: A 14-item questionnaire with 2 subscales: anxiety and depression. Each item is rated on a 4-point scale (0-3), giving maximum scores of 21 for anxiety and for depression. Scores of 11 or more on either subscale are considered to be a significant case of psychological morbidity, while scores of 8-10 represent 'borderline' and 0-7 represent 'normal.' Mixed-effects model repeated measures (MMRM) analysis was used to calculate Least Squares (LS) Mean and 95% Confidence Interval (CI). LS Mean values are controlled for treatment, site, baseline value, visit, treatment*visit and baseline*visit.
Time Frame: Baseline, Week 8
Population: All randomized participants who received at least one dose of study drug, and had baseline and at least one post-baseline HADS measurements during Weeks 1-8 (Study Period II).
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Duloxetine | Pregabalin
Number analyzed (Participants) | 399 | 402
units on a scale
  Anxiety Subscale Score (n= 398, 400) | -1.991 [-2.301 to -1.681] | -1.433 [-1.739 to -1.127]
  Depression Subscale Score | -1.064 [-1.351 to -0.778] | -0.642 [-0.925 to -0.359]
Statistical Analysis 1: Comparison: Duloxetine vs Pregabalin; Test type: Superiority or Other; p = 0.008, Mixed Models Analysis — P-value is for anxiety subscale score; LS Mean Difference (Final Values) = -0.558
Statistical Analysis 2: Comparison: Duloxetine vs Pregabalin; Test type: Superiority or Other; p = 0.031, Mixed Models Analysis — p-value is for depression subscale score; LS Mean Difference (Final Values) = -0.423

17. Secondary Outcome: Mean Change From Week 8 to Week 16 Endpoint in Hospital Anxiety and Depression Scale (HADS)
Description: A 14-item questionnaire with 2 subscales: anxiety and depression. Each item is rated on a 4-point scale (0-3), giving maximum scores of 21 for anxiety and for depression. Scores of 11 or more on either subscale are considered to be a significant case of psychological morbidity, while scores of 8-10 represent 'borderline' and 0-7 represent 'normal.' Mixed-effects model repeated measures (MMRM) analysis was used to calculate Least Squares (LS) Mean and 95% Confidence Interval (CI). LS Mean values are controlled for treatment, site, baseline value, visit, treatment*visit, baseline*visit and treatment in Study Period II.
Time Frame: Week 8, Week 16
Population: All randomized participants who received at least one dose of study drug, and had Week 8 and at least one HADS measurements during Weeks 9-16 (Study Period III).
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Combination | Monotherapy
Number analyzed (Participants) | 169 | 170
units on a scale
  Anxiety Subscale Score (n=169, 169) | -0.860 [-1.342 to -0.377] | -0.245 [-0.742 to 0.253]
  Depression Subscale Score (n=168, 170) | -0.461 [-0.916 to -0.007] | -0.083 [-0.550 to 0.384]
Statistical Analysis 1: Comparison: Combination vs Monotherapy; Test type: Superiority or Other; p = 0.049, Mixed Models Analysis — P-value is for anxiety subscale score; LS Mean Difference (Final Values) = -0.615
Statistical Analysis 2: Comparison: Combination vs Monotherapy; Test type: Superiority or Other; p = 0.198, Mixed Models Analysis — P-value is for depression subscale score; LS Mean Difference (Final Values) = -0.378

18. Other Pre Specified Outcome: Resource Utilization (Number of Days Hospitalized, Number of Days of Sick Leave) Baseline Through Week 8
Description: Data presented are the number of days hospitalized and work/school missed (sick leave) due to diabetic peripheral neuropathic pain (DPNP) during the last 8 weeks.
Time Frame: Baseline through Week 8
Population: All randomized participants who received at least one dose of study drug and provided information of hospitalization and sick leave during Weeks 1-8 (Study Period II).
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Duloxetine | Pregabalin
Number analyzed (Participants) | 314 | 319
days
  Days hospitalized | 0 (0.00) | 0 (0.00)
  Days of sick leave (n=108, 101) | 1.9 (8.34) | 0.3 (2.04)

19. Secondary Outcome: Resource Utilization (Number of Days Hospitalized, Number of Days of Sick Leave) Week 8 Through Week 16
Description: as for outcome 18
Time Frame: Week 8 through Week 16
Population: All randomized participants who received at least one dose of study drug and provided information of hospitalization and sick leave during Weeks 9-16 (Study Period III).
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Combination | Monotherapy
Number analyzed (Participants) | 140 | 146
days
  Days hospitalized (n=140, 146) | 0 (0.00) | 0 (0.00)
  Days of sick leave (n=41, 36) | 0.1 (0.65) | 0.4 (2.67)

20. Other Pre Specified Outcome: Average Number of Hours Worked for Pay Per Week Baseline Through Week 8
Description: Data presented are the average number of hours worked for pay per week during the last 8 weeks.
Time Frame: Baseline through Week 8
Population: All randomized participants who received at least one dose of study drug and had worked for pay during Weeks 1-8 (Study Period II).
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Duloxetine | Pregabalin
Number analyzed (Participants) | 102 | 100
hours | 37.6 (18.72) | 42.4 (15.52)

21. Other Pre Specified Outcome: Average Number of Hours Worked for Pay Per Week Week 8 Through Week 16
Description: Data presented are the average number of hours worked for pay per week during the last 8 weeks.
Time Frame: Week 8 through Week 16
Population: All randomized participants who received at least one dose of study drug and had worked for pay during Weeks 9-16 (Study Period III).
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Combination | Monotherapy
Number analyzed (Participants) | 42 | 36
hours | 39.8 (15.98) | 34.7 (21.46)

22. Other Pre Specified Outcome: Patient Global Impression of Improvement (PGI-I) Score at Week 8 Endpoint
Description: Measures participant's perception of improvement at the time of assessment compared with the start of treatment. The score ranges from 1 (very much better) to 7 (very much worse). Mixed-effects model repeated measures (MMRM) analysis was used to calculate Least Squares (LS) Mean and 95% Confidence Interval (CI). LS Mean values are controlled for treatment, site, visit, and treatment*visit.
Time Frame: Week 8
Population: All randomized participants who received at least one dose of study drug, and at least one post-baseline PGI-I measurement during Weeks 1-8 (Study Period II).
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Duloxetine | Pregabalin
Number analyzed (Participants) | 401 | 403
units on a scale | 2.601 [2.477 to 2.725] | 2.944 [2.821 to 3.067]
Statistical Analysis 1: Comparison: Duloxetine vs Pregabalin; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; LS Mean Difference (Final Values) = -0.343

23. Secondary Outcome: Patient Global Impression of Improvement (PGI-I) Score at Week 16 Endpoint
Description: Measures participant's perception of improvement at the time of assessment compared with the start of treatment for Study Period III. The score ranges from 1 (very much better) to 7 (very much worse). Mixed-effects model repeated measures (MMRM) analysis was used to calculate Least Squares (LS) Mean and 95% Confidence Interval (CI). LS Mean values are controlled for treatment, site, baseline value, visit, treatment*visit, baseline*visit and treatment in Study Period II.
Time Frame: Week 16
Population: All randomized participants who received at least one dose of study drug, and at least one PGI-I measurement during Weeks 9-16 (Study Period III).
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Combination | Monotherapy
Number analyzed (Participants) | 169 | 170
units on a scale | 2.256 [2.085 to 2.426] | 2.350 [2.174 to 2.526]
Statistical Analysis 1: Comparison: Combination vs Monotherapy; Test type: Superiority or Other; p = 0.385, Mixed Models Analysis; LS Mean Difference (Final Values) = -0.095

24. Other Pre Specified Outcome: Mean Change in Blood Pressure (BP) From Baseline to Week 8 Endpoint
Description: Least Squares (LS) mean values are controlled for treatment, site, baseline value, and treatment*site.
Time Frame: Baseline, Week 8
Population: All randomized participants who received at least one dose of study drug, and had baseline and at least one post-baseline BP measurement during Week 1-8 (Study Period II). Last observation carried forward (LOCF) principle was used.
Measure: Least Squares Mean (95% Confidence Interval); unit: millimeter of mercury (mm Hg)
Arm/Group | Duloxetine | Pregabalin
Number analyzed (Participants) | 386 | 389
millimeter of mercury (mm Hg)
  Systolic BP | -3.702 [-5.216 to -2.188] | -1.682 [-3.191 to -0.174]
  Diastolic BP | -0.816 [-1.766 to 0.134] | -0.951 [-1.898 to -0.003]
Statistical Analysis 1: Comparison: Duloxetine vs Pregabalin; Test type: Superiority or Other; p = 0.064, ANCOVA — P-value is for systolic BP; LS Mean Difference (Final Values) = -2.020
Statistical Analysis 2: Comparison: Duloxetine vs Pregabalin; Test type: Superiority or Other; p = 0.843, ANCOVA — P-value is for diastolic BP; LS Mean Difference (Final Values) = 0.135

25. Secondary Outcome: Mean Change in Blood Pressure (BP) From Week 8 to Week 16 Endpoint
Description: Least Squares (LS) mean values are controlled for treatment, site, baseline value, treatment*site and treatment in Study Period II.
Time Frame: Week 8, Week 16
Population: All randomized participants who received at least one dose of study drug, and had Week 8 and at least one BP measurement during Weeks 9-16 (Study Period III). Last observation carried forward (LOCF) principle was used.
Measure: Least Squares Mean (95% Confidence Interval); unit: millimeter of mercury (mm Hg)
Arm/Group | Combination | Monotherapy
Number analyzed (Participants) | 169 | 168
millimeter of mercury (mm Hg)
  Systolic BP | -1.206 [-3.202 to 0.790] | 0.124 [-1.891 to 2.138]
  Diastolic BP | -0.555 [-1.865 to 0.755] | -0.551 [-1.873 to 0.771]
Statistical Analysis 1: Comparison: Combination vs Monotherapy; Test type: Superiority or Other; p = 0.354, ANCOVA — P-value is for systolic BP; LS Mean Difference (Final Values) = -1.329
Statistical Analysis 2: Comparison: Combination vs Monotherapy; Test type: Superiority or Other; p = 0.997, ANCOVA — P-value is for diastolic BP; LS Mean Difference (Final Values) = -0.003

26. Other Pre Specified Outcome: Mean Change in Heart Rate From Baseline to Week 8 Endpoint
Description: Least Squares (LS) mean values are controlled for treatment, site, baseline value, and treatment*site.
Time Frame: Baseline, Week 8
Population: All randomized participants who received at least one dose of study drug, and had baseline and at least one post-baseline heart rate measurement during Weeks 1-8 (Study Period II). Last observation carried forward (LOCF) principle was used.
Measure: Least Squares Mean (95% Confidence Interval); unit: beats per minute (bpm)
Arm/Group | Duloxetine | Pregabalin
Number analyzed (Participants) | 384 | 389
beats per minute (bpm) | 0.839 [-0.062 to 1.741] | -2.478 [-3.369 to -1.588]
Statistical Analysis 1: Comparison: Duloxetine vs Pregabalin; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference (Final Values) = 3.317

27. Secondary Outcome: Mean Change in Heart Rate From Week 8 to Week 16 Endpoint
Description: as for outcome 25
Time Frame: Week 8, Week 16
Population: All randomized participants who received at least one dose of study drug, and had Week 8 and at least one heart rate measurement during Weeks 9- 16 (Study Period III). Last observation carried forward (LOCF) principle was used.
Measure: Least Squares Mean (95% Confidence Interval); unit: beats per minute (bpm)
Arm/Group | Combination | Monotherapy
Number analyzed (Participants) | 169 | 168
beats per minute (bpm) | 1.025 [-0.326 to 2.376] | 1.968 [0.602 to 3.333]
Statistical Analysis 1: Comparison: Combination vs Monotherapy; Test type: Superiority or Other; p = 0.332, ANCOVA; LS Mean Difference (Final Values) = -0.942

28. Other Pre Specified Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAE) Between Baseline and Week 8 Endpoint
Description: TEAEs in Study Period II are events that began or worsened after Week 0 compared with the period before Week 0.
Time Frame: Baseline through Week 8
Population: All randomized participants who received at least one dose of study drug during Weeks 1-8 (Study Period II).
Measure: Number; unit: participants
Arm/Group | Duloxetine | Pregabalin
Number analyzed (Participants) | 401 | 403
participants | 223 | 232
Statistical Analysis 1: Comparison: Duloxetine vs Pregabalin; Test type: Superiority or Other; p = 0.618, Fisher Exact

29. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) Between Week 8 and Week 16 Endpoint
Description: TEAEs in Study Period III are events that began or worsened after Week 8 compared with the period before Week 8.
Time Frame: Week 8 through Week 16
Population: All randomized participants who received at least one dose of study drug during Weeks 9-16 (Study Period III).
Measure: Number; unit: participants
Arm/Group | Combination | Monotherapy
Number analyzed (Participants) | 169 | 170
participants | 62 | 57
Statistical Analysis 1: Comparison: Combination vs Monotherapy; Test type: Superiority or Other; p = 0.571, Fisher Exact

30. Other Pre Specified Outcome: Number of Participants Who Discontinued From Study Between Baseline and Week 8 Endpoint
Time Frame: Baseline through Week 8
Population: All randomized participants who received at least one dose of study drug during Weeks 1-8 (Study Period II).
Measure: Number; unit: participants
Arm/Group | Duloxetine | Pregabalin
Number analyzed (Participants) | 401 | 403
participants | 68 | 70
Statistical Analysis 1: Comparison: Duloxetine vs Pregabalin; Test type: Superiority or Other; p = 0.744, Fisher Exact

31. Secondary Outcome: Number of Participants Who Discontinued From Study Between Week 8 and Week 16 Endpoint
Time Frame: Week 8 through Week 16
Population: All randomized participants who received at least one dose of study drug during Weeks 9-16 (Study Period III).
Measure: Number; unit: participants
Arm/Group | Combination | Monotherapy
Number analyzed (Participants) | 169 | 170
participants | 21 | 21
Statistical Analysis 1: Comparison: Combination vs Monotherapy; Test type: Superiority or Other; p = 1.000, Fisher Exact

ADVERSE EVENTS:
Arm/Group | Duloxetine (SP II) | Pregabalin (SP II) | Duloxetine (SP III) | DLX + PGB (SP III) | PGB + DLX (SP III) | Pregabalin (SP III)
Serious Adverse Events (participants affected / at risk) | 12/401 | 13/403 | 3/73 | 3/75 | 5/94 | 2/97
Other Adverse Events (participants affected / at risk) | 216/401 | 225/403 | 18/73 | 21/75 | 39/94 | 37/97
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Duloxetine (SP II) (N=401) | Pregabalin (SP II) (N=403) | Duloxetine (SP III) (N=73) | DLX + PGB (SP III) (N=75) | PGB + DLX (SP III) (N=94) | Pregabalin (SP III) (N=97)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Duodenitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hernia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchopneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pilonidal cyst (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Brain contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatitis c antibody positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myelitis transverse (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disorientation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hallucination (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Duloxetine (SP II) (N=401) | Pregabalin (SP II) (N=403) | Duloxetine (SP III) (N=73) | DLX + PGB (SP III) (N=75) | PGB + DLX (SP III) (N=94) | Pregabalin (SP III) (N=97)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 4 (4) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 8 (8) | 26 (27) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eyelid oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 5 (6) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Visual impairment (Eye disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 5 (5) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aphthous stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chapped lips (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 16 (17) | 13 (14) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 14 (14) | 11 (12) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Dry mouth (Gastrointestinal disorders) | 16 (17) | 9 (11) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 4 (4) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 4 (4) | 5 (5) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 5 (5) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 57 (61) | 25 (26) | 2 (2) | 1 (1) | 4 (4) | 1 (1)
Paraesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 12 (13) | 6 (7) | 0 (0) | 0 (0) | 4 (4) | 1 (1)
Asthenia (General disorders) | 6 (8) | 7 (7) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Discomfort (General disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Facial pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 18 (18) | 13 (13) | 2 (2) | 1 (1) | 2 (2) | 1 (1)
Gait disturbance (General disorders) | 1 (1) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema (General disorders) | 1 (1) | 7 (7) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 4 (5) | 21 (23) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pain (General disorders) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Therapeutic response unexpected (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 3 (3) | 5 (5) | 0 (0) | 0 (0) | 2 (3) | 1 (1)
Onychomycosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vaginal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Visual acuity tests abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vitamin b12 decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight increased (Investigations) | 2 (2) | 9 (9) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 17 (18) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 4 (7) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Increased appetite (Metabolism and nutrition disorders) | 0 (0) | 6 (6) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (4) | 4 (4) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 5 (6) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Muscle contracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 (5) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (4) | 3 (3) | 3 (3) | 2 (3) | 0 (0)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Amnesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Balance disorder (Nervous system disorders) | 4 (5) | 7 (7) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Disturbance in attention (Nervous system disorders) | 2 (2) | 7 (8) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Dizziness (Nervous system disorders) | 29 (36) | 61 (69) | 4 (5) | 2 (2) | 2 (2) | 2 (2)
Dysaesthesia (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dysarthria (Nervous system disorders) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 19 (21) | 13 (15) | 3 (3) | 0 (0) | 1 (4) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hypotonia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 7 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine with aura (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Paraesthesia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Psychomotor skills impaired (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sedation (Nervous system disorders) | 3 (3) | 3 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sensory loss (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 40 (46) | 44 (50) | 1 (1) | 0 (0) | 2 (2) | 5 (5)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Apathy (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 4 (6) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dissociation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 8 (8) | 4 (4) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Libido decreased (Psychiatric disorders) | 2 (2) | 5 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Loss of libido (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Mood swings (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paranoia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Restlessness (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sleep disorder (Psychiatric disorders) | 6 (6) | 6 (6) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dysuria (Renal and urinary disorders) | 9 (9) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Urinary hesitation (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urine flow decreased (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 6 (6) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 16 (16) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (2) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3)
Arteriosclerosis (Vascular disorders) | 3 (3) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 7 (7) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombophlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Venous insufficiency (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days